CLINICAL TRIAL: NCT01284335
Title: A Phase 1 Multicenter, Dose-escalation Study of LY573636-sodium in Combination With 1) Gemcitabine HCl or 2) Docetaxel or 3) Temozolomide or 4) Cisplatin, or 5) Erlotinib in Patients With Advanced Solid Tumors
Brief Title: A Safety Study in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to the termination of tasisulam development.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12267; H8K-MC-JZAK (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-19; First posted 2011-01-27 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors; Unresectable; Metastatic; Limited treatment options; Measurable or nonmeasurable disease
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Gemcitabine; Docetaxel; Temozolomide; Cisplatin; Erlotinib Hydrochloride; N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Gemcitabine plus LY573636 (Experimental)
  Interventions: Drug: Gemcitabine; Drug: LY573636
- Docetaxel plus LY573636 (Experimental)
  Interventions: Drug: Docetaxel; Drug: LY573636
- Temozolomide plus LY573636 (Experimental)
  Interventions: Drug: Temozolomide; Drug: LY573636
- Cisplatin plus LY573636 (Experimental)
  Interventions: Drug: Cisplatin; Drug: LY573636
- Erlotinib plus LY573636 (Experimental)
  Interventions: Drug: Erlotinib; Drug: LY573636

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 administered intravenously on Days 1 and 15 of a 28 day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Other Names: LY18011
  Arms: Gemcitabine plus LY573636
Drug: Docetaxel — 60 mg/m2 administered intravenously over 60 minutes on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Arms: Docetaxel plus LY573636
Drug: Temozolomide — 200 mg/m2 administered orally on days 1-5 of a 28 day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Arms: Temozolomide plus LY573636
Drug: Cisplatin — 75 mg/m2 administered intravenously on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Arms: Cisplatin plus LY573636
Drug: Erlotinib — 150 mg administered orally days 1-28 of a 28 day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Arms: Erlotinib plus LY573636
Drug: LY573636 — Individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Other Names: Tasisulam; LY573636-sodium

SUMMARY:
The purpose of this study is to determine a safe dose of LY573636 (tasisulam) when used in 5 separate combinations with an approved cancer medication for treating participants with advanced cancer. Data from this study will be reviewed for any side effects or anti-tumor activity that may be associated with the LY573636 combination treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have histologically confirmed solid malignancy or lymphoma that is unresectable and/or metastatic for which monotherapy with gemcitabine HCl, docetaxel, temozolomide, cisplatin, or erlotinib would otherwise be appropriate
* Must have tumor progression after receiving standard/approved chemotherapy or limited treatment options
* Must have measurable or nonmeasurable disease
* Have given written informed consent prior to any study-specific procedures
* Must have adequate hepatic, hematologic and renal function
* Must have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy or other investigational therapy for at least 4 weeks (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy. Endocrine therapies for the treatment of prostate cancer may be continued, at the discretion of the investigator. Whole brain radiation must have been completed 90 days before starting study therapy. Participants without evidence of brain metastases who have received prophylactic whole brain irradiation as part of standard of care for small cell lung cancer may be included in the study with a shorter washout period pending approval by the Lilly physician.
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 6 months following the last dose of study drug.
* Females with child-bearing potential must have had a negative serum pregnancy test within 7 days prior to the first dose of study drug.
* Must have a serum albumin level greater than or equal to 3.0 g/dL (30 g/L).
* Must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale

Exclusion Criteria:

* Have received treatment within 30 days of the initial dose of study drug with a drug that has not received regulatory approval for any indication
* Have serious preexisting medical conditions that in the opinion of the investigator would preclude participation in the study
* Participants with active central nervous system or brain metastasis at the time of study entry. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before study entry to rule out brain metastasis. Participants with stable CNS metastasis not requiring steroids may be eligible.
* Have a current hematologic malignancy (other than lymphoma)
* Participants with serious concomitant disorders, including active bacterial, fungal, or viral infection, incompatible with the study)
* Participants actively receiving warfarin (Coumadin®) therapy
* Participants who have previously completed or withdrawn from any study investigating LY573636
* Participants with a known hypersensitivity to one of the combination drugs cannot be enrolled to the treatment arm which includes that chemotherapeutic combination
* Females who are pregnant or breast feeding
* Have known positive test results of HIV, hepatitis B, or hepatitis C
* Participants receiving amiodarone, quinidine, propofol, or clozapine.
* Participants receiving treatment with strong or moderate inhibitors of CYP2C19, including proton-pump inhibitors (PPIs). Esomeprazole or pantoprazole are allowed if not administered 72 hours before or after LY573636 administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2008-07; Primary Completion 2012-10 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 or Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- United States (19):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fayetteville, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Park Ridge, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kettering, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Woodlands, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tyler, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yakima, Washington

REFERENCES:
- [Derived] Jotte RM, Von Hoff DD, Braiteh F, Becerra CR, Richards DA, Smith DA, Garbo L, Stephenson J, Conkling PR, Robert-Vizcarrondo F, Chen J, Turner PK, Chow KH, Tai DF, Ilaria R Jr. An innovative, multi-arm, complete phase 1b study of the novel anti-cancer agent tasisulam in patients with advanced solid tumors. Invest New Drugs. 2015 Feb;33(1):148-58. doi: 10.1007/s10637-014-0160-z. Epub 2014 Sep 28. PMID 25260842

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study completion was defined as when the recommended dose of LY573636 (tasisulam) was defined for each treatment arm or if a decision was made to stop enrollment in the study for business reasons.
Groups:
- Arm A Tasisulam + Gemcitabine Dose Escalation; Arm A Tasisulam + Gemcitabine Dose Confirmation: Gemcitabine 1000 milligrams meter squared (mg/m2) administered intravenously on Days 1 and 15 of a 28 day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Tasisulam dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
- Arm B* Tasisulam + Docetaxel Dose Escalation: Tasisulam and Docetaxel 60 mg/m2 administered concurrently intravenously on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
- Arm B1 Tasisulam + Docetaxel Dose Escalation: Docetaxel 60 mg/m2 administered intravenously over 60 minutes on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Tasisulam Day 4 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
- Arm B2 Tasisulam + Docetaxel Dose Escalation; Arm B2 Tasisulam + Docetaxel Dose Confirmation: Tasisulam individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Docetaxel 60 mg/m2 administered intravenously over 60 minutes on Day 4 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
- Arm C Tasisulam + Temozolomide Dose Escalation; Arm C Tasisulam + Temozolomide Dose Confirmation: Tasisulam individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Temozolomide 200 mg/m2 administered orally on days 1-5 of a 28 day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met
- Arm D* Tasisulam + Cisplatin Dose Escalation: Tasisulam and 75 mg/m2 cisplatin administered IV on Day 1 in 21-day cycles.
- Arm D Tasisulam + Cisplatin Dose Escalation; Arm D Tasisulam + Cisplatin Dose Confirmation: Tasisulam individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Cisplatin 75 mg/m2 administered intravenously on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
- Arm E Tasisulam + Erlotinib Dose Escalation; Arm E Tasisulam + Erlotinib Dose Confirmation: Tasisulam individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Erlotinib 150 mg administered orally (PO) days 1-28 of a 28 day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
Period: Overall Study
Arm/Group | Arm A Tasisulam + Gemcitabine Dose Escalation | Arm A Tasisulam + Gemcitabine Dose Confirmation | Arm B* Tasisulam + Docetaxel Dose Escalation | Arm B1 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Confirmation | Arm C Tasisulam + Temozolomide Dose Escalation | Arm C Tasisulam + Temozolomide Dose Confirmation | Arm D* Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Confirmation | Arm E Tasisulam + Erlotinib Dose Escalation | Arm E Tasisulam + Erlotinib Dose Confirmation
Started | 25 | 33 | 5 | 5 | 24 | 26 | 19 | 6 | 4 | 14 | 45 | 16 | 12
Received at Least One Dose of Study Drug | 25 | 33 | 5 | 5 | 24 | 26 | 19 | 6 | 4 | 14 | 45 | 16 | 12
Completed | 25 | 33 | 5 | 5 | 24 | 26 | 19 | 6 | 4 | 14 | 45 | 16 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received at least one dose of study drug.
Groups:
- Arm B1 Tasisulam + Docetaxel Dose Escalation: Docetaxel 60 mg/m2 administered intravenously over 60 minutes on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Tasisulam Day 4 of a 28 day cycle. Participant's may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
- Total: Total of all reporting groups
Arm/Group | Arm A Tasisulam + Gemcitabine Dose Escalation | Arm A Tasisulam + Gemcitabine Dose Confirmation | Arm B* Tasisulam + Docetaxel Dose Escalation | Arm B1 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Confirmation | Arm C Tasisulam + Temozolomide Dose Escalation | Arm C Tasisulam + Temozolomide Dose Confirmation | Arm D* Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Confirmation | Arm E Tasisulam + Erlotinib Dose Escalation | Arm E Tasisulam + Erlotinib Dose Confirmation | Total
Number analyzed (Participants) | 25 | 33 | 5 | 5 | 24 | 26 | 19 | 6 | 4 | 14 | 45 | 16 | 12 | 234
Age, Continuous [Median (Full Range); unit: years] | 63.2 [56.6 to 81.5] | 65.5 [21.4 to 83.0] | 66.3 [54.2 to 77.3] | 78.8 [73.0 to 82.1] | 64.2 [37.1 to 83.2] | 62.7 [30.0 to 83.0] | 63.3 [31.0 to 78.3] | 65.7 [50.4 to 84.4] | 48.46 [39.22 to 67.27] | 54.88 [31.45 to 75.60] | 67.36 [30.53 to 89.50] | 57.84 [32.42 to 81.28] | 61.63 [52.07 to 78.16] | 63.6 [21.4 to 89.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 3 | 2 | 10 | 17 | 4 | 3 | 3 | 7 | 21 | 9 | 7 | 117
  Male | 13 | 14 | 2 | 3 | 14 | 9 | 15 | 3 | 1 | 7 | 24 | 7 | 5 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African | 1 | 2 | 1 | 2 | 2 | 3 | 0 | 0 | 0 | 2 | 6 | 3 | 0 | 22
  Race: Caucasian | 23 | 30 | 3 | 3 | 22 | 21 | 17 | 6 | 3 | 10 | 36 | 12 | 11 | 197
  Race: East Asian | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 7
  Race: West Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Race: Hispanic | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 33 | 5 | 5 | 24 | 26 | 19 | 6 | 4 | 14 | 45 | 16 | 12 | 234

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities Cycle 1
Description: A Dose-Limiting Toxicity (DLT) is defined as an Adverse Event (AE) that is likely related to the study medication or combination, and fulfills any one of the following criteria: Common Terminology Criteria for Adverse Events (CTCAE, Version 3.0) Grade 4 neutropenia lasting more than 5 days. Grade 4 neutropenia with fever or Grade 4 thrombocytopenia, regardless of duration; Grade ≥3 thrombocytopenia with bleeding, regardless of duration; Grade ≥3 nonhematologic toxicity (excluding nausea/vomiting or diarrhea that can be controlled with medication, and alopecia). Grade 3 electrolyte toxicity (for example, hypokalemia, hypophosphatemia) will not be considered a DLT unless it is considered related to the study drug or combination and does not resolve with standard replacement treatments within 42 days after Cycle 1 Day 1. A summary of other nonserious AEs and all Serious Adverse Events (SAE), regardless of causality is located in the Reported Adverse Event section.
Time Frame: Baseline to Cycle 1 (Up to Day 28)
Population: All participants who received at least one dose of study drug Tasisulam in dose escalation phase and experienced a dose-limiting toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Tasisulam + Gemcitabine Dose Escalation | Arm A Tasisulam + Gemcitabine Dose Confirmation | Arm B* Tasisulam + Docetaxel Dose Escalation | Arm B1 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Confirmation | Arm C Tasisulam + Temozolomide Dose Escalation | Arm C Tasisulam + Temozolomide Dose Confirmation | Arm D* Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Confirmation | Arm E Tasisulam + Erlotinib Dose Escalation | Arm E Tasisulam + Erlotinib Dose Confirmation
Number analyzed (Participants) | 25 | 33 | 5 | 5 | 24 | 26 | 19 | 6 | 4 | 14 | 45 | 16 | 12
Participants | 4 | 0 | 4 | 4 | 3 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 0

2. Secondary Outcome: Pharmacokinetic (PK): Concentration Maximum (Cmax)
Description: Cycle 2: predose,1h start of infusion, end of infusion, 30min,2h,4h,6h,22h,166h,334h,698h end of infusion.
Time Frame: Cycle 1: predose,0,30min,1h start of infusion, end of infusion, 30min,2h,4h,6h,22h,166h,334h,698h end of infusion.
Population: All participants who received at least one dose of study drug Tasisulam and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- Tasisulam: Tasisulam dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion are met.
Arm/Group | Tasisulam
Number analyzed (Participants) | 217
micrograms per milliliter (µg/mL)
  Cycle 1 | 306 (20.03)
  Cycle 2: number analyzed (Participants) | 159
  Cycle 2 | 250 (31.39)

3. Secondary Outcome: Percentage of Participants With a Complete (CR) or Partial Response (PR) (Best Overall Tumor Response)
Description: Best overall tumor response was evaluated using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.0) criteria. Complete Response (CR) was defined as the disappearance of all target lesions; Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to Study Completion (Up to 2 years)
Population: All participants who received study drug Tasisulam and had CR or PR tumor response at dose confirmation phase.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm B* Tasisulam + Docetaxel Dose Confirmation: Tasisulam and Docetaxel 60 mg/m2 administered concurrently intravenously on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
Arm/Group | Arm A Tasisulam + Gemcitabine Dose Confirmation | Arm B* Tasisulam + Docetaxel Dose Confirmation | Arm C Tasisulam + Temozolomide Dose Confirmation | Arm D Tasisulam + Cisplatin Dose Confirmation | Arm E Tasisulam + Erlotinib Dose Confirmation
Number analyzed (Participants) | 33 | 26 | 6 | 45 | 12
percentage of participants
  Non-Small Cell Lung Cancer (NSCLC): number analyzed (Participants) | 4 | 10 | 0 | 20 | 4
  Non-Small Cell Lung Cancer (NSCLC) | 0.0 [0 to 0] | 20.0 [3.7 to 50.7] |  | 5.0 [0.3 to 21.6] | 0.0 [0 to 0]
  Other: number analyzed (Participants) | 14 | 16 | 6 | 10 | 7
  Other | 14.3 [2.6 to 38.5] | 6.3 [0.3 to 26.4] | 0.0 [0 to 0] | 10.0 [0.5 to 39.4] | 14.3 [0.7 to 52.1]
  Pancreas: number analyzed (Participants) | 15 | 0 | 0 | 1 | 1
  Pancreas | 13.3 [2.4 to 36.3] |  |  | 0 [0.0 to 0.0] | 0.0 [0 to 0]
  Small Cell Lung Cancer (SCLC): number analyzed (Participants) | 0 | 0 | 0 | 14 | 0
  Small Cell Lung Cancer (SCLC) |  |  |  | 7.1 [0.4 to 29.7] |

4. Secondary Outcome: Number of Participants With a Clinically Significant Effects
Description: Clinically significant effects are reported if a Grade 3 or higher treatment emergent adverse event (TEAE) and observed in ≥10% of participants or a toxicity possibly related to study drug based on Common Terminology Criteria for Adverse Events (CTCAE). A summary of other nonserious AEs and all SAEs, regardless of causality is located in the Reported Adverse Event section.
Time Frame: Baseline to Study Completion (Up to 2 years)
Population: All participants who received at least one dose of study drug Tasisulam and experienced a Grade 3 or higher TEAE or drug toxicity possibly related to study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A Tasisulam + Gemcitabine Dose Escalation; Arm A Tasisulam + Gemcitabine Dose Confirmation: Gemcitabine 1000 milligrams meter squared (mg/m2) administered intravenously on Days 1 and 15 of a 28 day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Tasisulam dose is dependent on participants height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
- Arm B1 Tasisulam + Docetaxel Dose Escalation; Arm B2 Tasisulam + Docetaxel Dose Escalation; Arm B2 Tasisulam + Docetaxel Dose Confirmation: Tasisulam individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Docetaxel 60 mg/m2 administered intravenously over 60 minutes on Day 4 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
Arm/Group | Arm A Tasisulam + Gemcitabine Dose Escalation | Arm A Tasisulam + Gemcitabine Dose Confirmation | Arm B1 Tasisulam + Docetaxel Dose Escalation | Arm B* Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Confirmation | Arm C Tasisulam + Temozolomide Dose Escalation | Arm C Tasisulam + Temozolomide Dose Confirmation | Arm D* Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam + Cisplatin Dose Confirmation | Arm E Tasisulam + Erlotinib Dose Escalation | Arm E Tasisulam + Erlotinib Dose Confirmation
Number analyzed (Participants) | 25 | 33 | 5 | 5 | 24 | 26 | 19 | 6 | 4 | 14 | 45 | 16 | 12
Participants
  TEAE >/= Grade 3 | 15 | 18 | 0 | 0 | 16 | 19 | 11 | 6 | 0 | 8 | 30 | 5 | 7
  Toxicity >/= Grade 3 | 13 | 18 | 5 | 4 | 18 | 26 | 13 | 6 | 1 | 7 | 30 | 5 | 7

5. Secondary Outcome: PK: Area Under the Curve Albumin (AUCalb)
Description: Cycle 2: predose,1h start of infusion, end of infusion, 30min,2h,4h,6h,22h,166h,334h,698h end of infusion.
Time Frame: Cycle 1: predose,0,30min,1h start of infusion, end of infusion, 30min,2h,4h,6h,22h,166h,334h,698h end of infusion.
Population: All participants who received at least one dose of study drug Tasisulam and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (µg*h/mL)
Groups:
- Tasisulam: Tasisulam dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters
Arm/Group | Tasisulam
Number analyzed (Participants) | 217
micrograms*hour/milliliter (µg*h/mL)
  Cycle 1 | 946 (427.2)
  Cycle 2: number analyzed (Participants) | 162
  Cycle 2 | 648 (765.92)

ADVERSE EVENTS:
Groups:
- Arm D Tasisulam+ Cisplatin Dose Escalation; Arm D Tasisulam+ Cisplatin Dose Confirmation: Tasisulam individualized dose is dependent on participant's height, weight, gender and is adjusted to target a specific exposure range corrected for a participant's laboratory parameters. Intravenous dosing is done on Day 1 of a 28 day cycle. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria are met.
  Cisplatin 75 mg/m2 administered intravenously on Day 1 of the 28-day cycle until disease progression, unacceptable toxicity or other discontinuation criteria are met.
Arm/Group | Arm A Tasisulam + Gemcitabine Dose Escalation | Arm A Tasisulam + Gemcitabine Dose Confirmation | Arm B* Tasisulam + Docetaxel Dose Escalation | Arm B1 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Escalation | Arm B2 Tasisulam + Docetaxel Dose Confirmation | Arm C Tasisulam + Temozolomide Dose Escalation | Arm C Tasisulam + Temozolomide Dose Confirmation | Arm D* Tasisulam + Cisplatin Dose Escalation | Arm D Tasisulam+ Cisplatin Dose Escalation | Arm D Tasisulam+ Cisplatin Dose Confirmation | Arm E Tasisulam + Erlotinib Dose Escalation | Arm E Tasisulam + Erlotinib Dose Confirmation
All-Cause Mortality (participants affected / at risk) | 2/25 | 8/33 | 1/5 | 1/5 | 0/24 | 4/26 | 3/19 | 3/6 | 1/4 | 2/14 | 7/45 | 3/16 | 3/12
Serious Adverse Events (participants affected / at risk) | 9/25 | 14/33 | 1/5 | 2/5 | 9/24 | 12/26 | 8/19 | 4/6 | 1/4 | 4/14 | 19/45 | 6/16 | 7/12
Other Adverse Events (participants affected / at risk) | 24/25 | 33/33 | 5/5 | 5/5 | 24/24 | 26/26 | 19/19 | 6/6 | 4/4 | 14/14 | 43/45 | 16/16 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A Tasisulam + Gemcitabine Dose Escalation (N=25) | Arm A Tasisulam + Gemcitabine Dose Confirmation (N=33) | Arm B* Tasisulam + Docetaxel Dose Escalation (N=5) | Arm B1 Tasisulam + Docetaxel Dose Escalation (N=5) | Arm B2 Tasisulam + Docetaxel Dose Escalation (N=24) | Arm B2 Tasisulam + Docetaxel Dose Confirmation (N=26) | Arm C Tasisulam + Temozolomide Dose Escalation (N=19) | Arm C Tasisulam + Temozolomide Dose Confirmation (N=6) | Arm D* Tasisulam + Cisplatin Dose Escalation (N=4) | Arm D Tasisulam+ Cisplatin Dose Escalation (N=14) | Arm D Tasisulam+ Cisplatin Dose Confirmation (N=45) | Arm E Tasisulam + Erlotinib Dose Escalation (N=16) | Arm E Tasisulam + Erlotinib Dose Confirmation (N=12)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 2 (3) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0/13 (0) | 1/14 (2) | 0/2 (0) | 0/3 (0) | 0/14 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0) | 0/1 (0) | 0/7 (0) | 0/24 (0) | 0/7 (0) | 0/5 (0)
Adrenal haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jejunal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm A Tasisulam + Gemcitabine Dose Escalation (N=25) | Arm A Tasisulam + Gemcitabine Dose Confirmation (N=33) | Arm B* Tasisulam + Docetaxel Dose Escalation (N=5) | Arm B1 Tasisulam + Docetaxel Dose Escalation (N=5) | Arm B2 Tasisulam + Docetaxel Dose Escalation (N=24) | Arm B2 Tasisulam + Docetaxel Dose Confirmation (N=26) | Arm C Tasisulam + Temozolomide Dose Escalation (N=19) | Arm C Tasisulam + Temozolomide Dose Confirmation (N=6) | Arm D* Tasisulam + Cisplatin Dose Escalation (N=4) | Arm D Tasisulam+ Cisplatin Dose Escalation (N=14) | Arm D Tasisulam+ Cisplatin Dose Confirmation (N=45) | Arm E Tasisulam + Erlotinib Dose Escalation (N=16) | Arm E Tasisulam + Erlotinib Dose Confirmation (N=12)
Anaemia (Blood and lymphatic system disorders) | 11 (66) | 13 (28) | 3 (5) | 4 (11) | 11 (45) | 11 (82) | 6 (21) | 2 (4) | 0 (0) | 5 (13) | 19 (71) | 8 (27) | 4 (14)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (11) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 4 (7) | 2 (4) | 1 (1) | 0 (0) | 1 (4) | 4 (12) | 0 (0) | 2 (5)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 13 (48) | 7 (30) | 4 (5) | 3 (17) | 14 (59) | 17 (84) | 6 (16) | 2 (3) | 1 (10) | 5 (24) | 19 (64) | 2 (6) | 5 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (41) | 11 (28) | 1 (1) | 0 (0) | 5 (7) | 11 (30) | 8 (33) | 4 (8) | 0 (0) | 6 (14) | 26 (89) | 4 (7) | 4 (24)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 3 (4) | 2 (11) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 4 (4) | 2 (2) | 1 (2)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (13) | 2 (7) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (22) | 4 (8) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 1 (2) | 0 (0)
Chorioretinal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (14) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (9) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (9) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 1 (6)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Abdominal hernia (Gastrointestinal disorders) | 1 (22) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (11) | 5 (9) | 0 (0) | 2 (4) | 3 (12) | 4 (15) | 2 (4) | 1 (2) | 2 (13) | 2 (6) | 3 (11) | 2 (5) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (2) | 3 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (26) | 16 (64) | 1 (7) | 2 (4) | 7 (24) | 13 (57) | 7 (25) | 2 (3) | 3 (6) | 4 (9) | 11 (48) | 3 (31) | 3 (15)
Diarrhoea (Gastrointestinal disorders) | 13 (22) | 9 (51) | 2 (4) | 4 (11) | 9 (18) | 7 (31) | 4 (6) | 1 (2) | 1 (1) | 1 (2) | 13 (99) | 10 (49) | 4 (20)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 2 (9)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 1 (8) | 1 (2) | 0 (0) | 1 (1) | 4 (17) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 2 (6) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (2) | 1 (5)
Flatulence (Gastrointestinal disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (11) | 0 (0) | 0 (0) | 0 (0) | 2 (43) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 1 (9) | 2 (5)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 2 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (50) | 7 (42) | 3 (3) | 3 (7) | 10 (21) | 10 (72) | 7 (22) | 0 (0) | 3 (20) | 4 (13) | 19 (126) | 6 (11) | 4 (6)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 3 (11) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (13) | 3 (4) | 2 (3) | 1 (2) | 7 (15) | 4 (14) | 4 (4) | 1 (1) | 1 (2) | 2 (6) | 15 (44) | 2 (3) | 6 (11)
Application site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 5 (12) | 4 (14) | 0 (0) | 0 (0) | 3 (9) | 1 (1) | 3 (7) | 0 (0) | 1 (2) | 0 (0) | 9 (78) | 2 (3) | 2 (4)
Chest discomfort (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 3 (3) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Decreased activity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (2) | 0 (0)
Fatigue (General disorders) | 17 (76) | 17 (90) | 3 (11) | 4 (8) | 16 (70) | 16 (97) | 13 (36) | 1 (2) | 3 (12) | 7 (37) | 27 (163) | 7 (26) | 5 (20)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 1 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 6 (11) | 4 (9) | 1 (3) | 1 (1) | 7 (20) | 4 (42) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (13) | 1 (8)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 2 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 4 (7) | 3 (13) | 2 (6) | 2 (3) | 5 (15) | 6 (100) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 6 (9) | 5 (13) | 1 (2)
Pain (General disorders) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 2 (9) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (6)
Pyrexia (General disorders) | 5 (5) | 5 (26) | 2 (5) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (3) | 3 (5) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (3)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 2 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Bronchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (5)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 1 (3)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (40) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (3) | 2 (5) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 3 (4) | 0 (0) | 0 (0) | 5 (10) | 1 (2) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (7) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/12 (0) | 0/19 (0) | 0/3 (0) | 0/2 (0) | 0/10 (0) | 0/17 (0) | 0/4 (0) | 0/3 (0) | 0/3 (0) | 0/7 (0) | 2/21 (3) | 0/9 (0) | 0/7 (0)
Vulvovaginitis (Infections and infestations) | 0/12 (0) | 1/19 (1) | 0/3 (0) | 0/2 (0) | 0/10 (0) | 0/17 (0) | 0/4 (0) | 0/3 (0) | 0/3 (0) | 0/7 (0) | 0/21 (0) | 0/9 (0) | 0/7 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 3 (9) | 3 (5) | 2 (2) | 0 (0) | 4 (15) | 1 (1) | 2 (12) | 1 (1) | 0 (0) | 3 (13) | 12 (66) | 0 (0) | 3 (10)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbon dioxide decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Precancerous cells present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 5 (13) | 5 (17) | 0 (0) | 0 (0) | 4 (7) | 1 (8) | 2 (5) | 1 (2) | 0 (0) | 2 (5) | 4 (8) | 3 (6) | 1 (2)
Weight increased (Investigations) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (22) | 6 (27) | 0 (0) | 2 (6) | 8 (23) | 8 (30) | 6 (19) | 2 (2) | 2 (5) | 3 (14) | 15 (36) | 9 (24) | 5 (14)
Dehydration (Metabolism and nutrition disorders) | 4 (10) | 2 (2) | 1 (1) | 0 (0) | 6 (7) | 3 (10) | 3 (3) | 0 (0) | 0 (0) | 3 (6) | 6 (10) | 2 (4) | 4 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (5) | 2 (6) | 0 (0) | 1 (7) | 2 (2) | 3 (5) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (9) | 6 (13) | 0 (0) | 2 (5) | 5 (11) | 9 (66) | 0 (0) | 1 (2) | 0 (0) | 4 (15) | 11 (22) | 6 (13) | 3 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (11) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (13) | 4 (15) | 1 (1) | 1 (2) | 6 (17) | 9 (26) | 1 (1) | 0 (0) | 1 (1) | 3 (10) | 12 (25) | 8 (19) | 5 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 4 (7) | 5 (7) | 4 (19) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 9 (10) | 1 (1) | 3 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 3 (4) | 0 (0) | 0 (0) | 2 (8) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 7 (9) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (11) | 3 (5) | 0 (0) | 4 (8) | 7 (24) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 10 (17) | 2 (3) | 3 (4)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (23) | 1 (9) | 1 (3) | 0 (0) | 4 (9) | 2 (9) | 1 (14) | 0 (0) | 1 (6) | 1 (10) | 2 (4) | 1 (2) | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (14) | 4 (5) | 0 (0) | 0 (0) | 2 (13) | 6 (13) | 0 (0) | 0 (0) | 1 (6) | 2 (20) | 4 (12) | 2 (4) | 2 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (19) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (70) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 1 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 1 (2) | 1 (7) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (3) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (10) | 1 (7) | 1 (3) | 0 (0) | 2 (7) | 2 (8) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (19) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (8) | 1 (2) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (8) | 1 (3) | 1 (9)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 3 (4) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 6 (50) | 0 (0) | 6 (33)
Dysgeusia (Nervous system disorders) | 2 (4) | 8 (37) | 0 (0) | 1 (2) | 4 (18) | 2 (8) | 3 (7) | 1 (1) | 1 (4) | 2 (8) | 5 (17) | 1 (2) | 2 (7)
Headache (Nervous system disorders) | 3 (13) | 2 (2) | 4 (5) | 0 (0) | 3 (4) | 3 (13) | 3 (8) | 1 (2) | 1 (6) | 0 (0) | 3 (4) | 0 (0) | 3 (16)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Neuropathy peripheral (Nervous system disorders) | 3 (7) | 2 (18) | 1 (1) | 1 (2) | 3 (7) | 4 (62) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 3 (11) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (24) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (6) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (9) | 0 (0) | 1 (3) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (22) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (14) | 0 (0) | 0 (0) | 2 (4) | 4 (10) | 0 (0) | 3 (5) | 1 (2) | 3 (6) | 3 (5) | 2 (41) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (7) | 2 (11) | 0 (0) | 0 (0) | 1 (12) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 1 (4) | 1 (3) | 3 (7) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (14) | 2 (6) | 0 (0) | 1 (3) | 3 (14) | 6 (16) | 4 (11) | 0 (0) | 1 (2) | 1 (6) | 5 (22) | 3 (5) | 3 (22)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (5)
Hydronephrosis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/13 (0) | 2/14 (8) | 0/2 (0) | 0/3 (0) | 0/14 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0) | 0/1 (0) | 0/7 (0) | 0/24 (0) | 0/7 (0) | 0/5 (0)
Testicular pain (Reproductive system and breast disorders) | 1/13 (2) | 0/14 (0) | 0/2 (0) | 0/3 (0) | 0/14 (0) | 0/9 (0) | 0/15 (0) | 0/3 (0) | 0/1 (0) | 0/7 (0) | 0/24 (0) | 0/7 (0) | 0/5 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/12 (0) | 1/19 (2) | 0/3 (0) | 0/2 (0) | 0/10 (0) | 0/17 (0) | 1/4 (1) | 0/3 (0) | 0/3 (0) | 0/7 (0) | 0/21 (0) | 0/9 (0) | 0/7 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (11) | 11 (43) | 2 (5) | 0 (0) | 7 (22) | 4 (10) | 6 (13) | 1 (2) | 1 (4) | 2 (2) | 10 (39) | 0 (0) | 3 (12)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (29) | 9 (35) | 1 (3) | 2 (5) | 7 (20) | 8 (88) | 5 (7) | 1 (1) | 0 (0) | 2 (4) | 10 (21) | 4 (7) | 2 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (15) | 2 (5) | 1 (1) | 0 (0) | 2 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (6) | 1 (5) | 1 (14)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5) | 1 (3) | 0 (0) | 2 (11) | 4 (9) | 2 (9) | 1 (2) | 1 (11) | 0 (0) | 6 (6) | 2 (9) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (14) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (5) | 2 (11) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (13) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 2 (9) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (8) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 2 (13) | 1 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 1 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (10) | 6 (28) | 1 (6) | 2 (10) | 7 (43) | 8 (77) | 1 (2) | 2 (3) | 0 (0) | 1 (6) | 6 (26) | 0 (0) | 2 (11)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (25) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (9) | 0 (0) | 0 (0) | 2 (16) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 4 (19) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (14)
Hirsutism (Skin and subcutaneous tissue disorders) | 0/12 (0) | 0/19 (0) | 0/3 (0) | 0/2 (0) | 0/10 (0) | 0/17 (0) | 1/4 (3) | 0/3 (0) | 0/3 (0) | 0/7 (0) | 0/21 (0) | 0/9 (0) | 0/7 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 1 (8) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (6) | 1 (5)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (9) | 2 (8) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (8) | 2 (10) | 0 (0) | 0 (0) | 8 (17) | 2 (8) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (18) | 7 (45)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (13) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 3 (7) | 1 (2)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (6) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (17) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to termination of development of the tasisulam compound. All participants were considered to have completed the study upon the completion of one cycle of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days